CLINICAL TRIAL: NCT01780493
Title: The Long Term Follow-Up Results Of The Direct Nipple Ureteroneocystostomy Technique: A Prospective Study
Brief Title: The Long Term Follow-Up Results Of The Direct Nipple Ureteroneocystostomy Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Assistant Professor, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03.04.2007/172
Record Dates: First submitted 2013-01-22; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Vesicoureteral Reflux; Nipple Ureteroneocystostomy
Keywords: Nipple; Technique; Ureter; Vesicoureteral Reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux

ARMS (1):
- Direct Nipple Ureteroneocystostomy (Other)
  Interventions: Procedure: The Direct Nipple Ureteroneocystostomy Technique

INTERVENTIONS:
Procedure: The Direct Nipple Ureteroneocystostomy Technique

SUMMARY:
To evaluate the long term follow-up results of the direct nipple ureteroneocystostomy technique.

ELIGIBILITY:
Inclusion Criteria:

* Megaureter.
* Ligated Ureter during surgery.

Exclusion Criteria:

* Neurogenic bladder
* Surgical wound infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-03; Primary Completion 2008-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Inter-IVU image differences and DMSA uptakes | 3 month after surgery
  In cases attending regular follow-ups, preoperative and postoperative 1st year DMSA results and amount of pelvicaliceal dilatation in the IVU of the unit that underwent surgery were compared statistically (by counting the dots falling on the pelvis and calices using stereologic methods which use transparent acetates with 3-mm inter-grid distances. Inter-IVU image differences between IVUs taken at different centers were resolved by using the value found by counting the dots falling on the 4th lumbar vertebra in both films and proportioning the results with each other as the multiplier. Measurable values were expressed as means + standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical Faculty, Department of Urology, Kayseri, Turkey (Türkiye)